CLINICAL TRIAL: NCT00926965
Title: Tardive Dyskinesia and Cognitive Function
Acronym: TD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Yu-Li Veterans Hospital, Yu-Li Veterans Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TD; TD
Record Dates: First submitted 2008-03-02; First posted 2009-06-24 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Tardive Dyskinesia; Neurocognitive Function
Keywords: tardive dyskinesia; neurocognitive function
MeSH Terms: conditions — Tardive Dyskinesia | interventions — Amisulpride; Olanzapine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Olanzapine group (Experimental): randomized to Olanzapine group with dose range of 2.5-30mg/day
  Interventions: Drug: Olanzapine
- Amisulpiride group (Experimental): the subjects were randomized to the amisulpiride group with dose range of 100 to 800mg/day
  Interventions: Drug: amisulpride
- FGA group (Active Comparator): The subjects were randomized to maintain the conventional antipsychotics
  Interventions: Drug: Conventional antipsychotics

INTERVENTIONS:
Drug: amisulpride — amisulpride tablet 100-1200mg/day for 24 months
  Other Names: solian
  Arms: Amisulpiride group
Drug: Olanzapine — Olanzapine tablet 2.5 to 30 mg/day for 24 months
  Other Names: zyprexa
  Arms: Olanzapine group
Drug: Conventional antipsychotics — the subjects were randomized to the conventional antipsychotic group to maintain their original conventional antipsychotics
  Other Names: conventional antipsychotic
  Arms: FGA group

SUMMARY:
Previous researchers indicate that impaired cognitive flexibility was the primary factor distinguishing patients with from those without tardive dyskinesia (TD)1, and cognitive dysfunction correlates positively with the severity of TD2. Longitudinal data raised the possibility that the association between cognitive dysfunction and TD may reflect not organic vulnerability to but rather a state marker for this movement disorder as "tardive dementia"3. Atypical antipsychotic had been reported to alleviate the severity of TD4 and improved neurocognitive function separately5. But no researchers ever investigated the correlation of the two effects simultaneously. This randomized, single-blind and controlled study compared the effect of atypical antipsychotic on TD, neurocognitive function and associated factors for these changes.

DETAILED DESCRIPTION:
Eighty chronic schizophrenia inpatients who received conventional antipsychotics for more than one year, and met Schooler and Kane's criteria for persistent TD were enrolled in the study. The subjects were randomized to three groups: the olanzapine, amisulpride and FGA (first generation antipsychotic) controlled groups. Neurocognitive function were assessed using Wisconsin Card Sorting Test (WSCT) and Continuous Performance test (CPT) at baseline, 12th week and 24th week. Clinical successive ratings were performed with Brief psychiatric Rating Scale (BPRS), AIMS (Abnormal Involuntary Movement Rating Scale), Simpson-Angus Rating Scale (SAS), Udvalg for Kliniske Undersogelser side effect ratings (UKU) and Barnes akathesia scale (BAS).To evaluate the influences of prognostic factors on tardive dyskinesia and neurocognitive function and to control for all potential confounding variables, longitudinal analyses on the repeated measures data were conducted using generalized estimating equation models (GEE).

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia inpatients who received conventional antipsychotics for more than one year,
* those who met Schooler and Kane's criteria for persistent TD.

Exclusion Criteria:

* mental retardation,
* organic mental disorder,
* pregnancy and allergy to trial drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
change of Abnormal Involuntary movement scale(AIMS), Wisconsin Card Sorting Test (WSCT) and Continuous Performance test (CPT) | 24 months

SECONDARY OUTCOMES:
Brief psychiatric Rating Scale (BPRS), Simpson-Angus Rating Scale (SAS), Udvalg for Kliniske Undersogelser side effect ratings (UKU) and Barnes akathesia scale (BAS).body weight, porlactin, metabolic components | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ya Mei Bai, M.D.,Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Yu-Li Veternas Hospital, Hualien City, Taiwan